CLINICAL TRIAL: NCT00038272
Title: A Phase I/II Randomized, Double-Blind, Placebo-Controlled Pilot Study of Beta-D-2,6-diaminopurine Dioxolane (DAPD) Versus DAPD Plus Mycophenolate Mofetil (MMF) in Treatment-Experienced Subjects
Brief Title: A Study of DAPD Alone Versus DAPD Plus MMF for Treatment of HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5165; 10090 (Registry Identifier: DAIDS ES); ACTG A5165; AACTG A5165
Record Dates: First submitted 2002-05-29; First posted 2002-05-30 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Placebos; Drug Therapy, Combination; Anti-HIV Agents; Mycophenolate Mofetil; 2,6-diaminopurine dioxolane; Treatment Experienced; DAPD; MMF
MeSH Terms: conditions — HIV Infections | interventions — Mycophenolic Acid; amdoxovir

INTERVENTIONS:
Drug: Mycophenolate mofetil
Drug: Amdoxovir

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, and side effects of beta-D-2,6-diaminopurine dioxolane (DAPD) compared to DAPD plus mycophenolate mofetil (MMF) when these drugs are added to the anti-HIV treatment regimens of people infected with HIV.

Some studies have shown that DAPD and MMF can help fight HIV. However, neither DAPD nor MMF has been approved by the Food and Drug Administration for treating HIV infection. This study will help doctors decide if DAPD and MMF are good drugs for treating HIV.

DETAILED DESCRIPTION:
The antiretroviral potency of DAPD varies among antiretroviral-experienced patients. In vitro studies indicate that the potency of DAPD can be markedly increased by the addition of MMF. Preliminary data indicate that MMF is well tolerated in patients with advanced HIV-1 disease. However, there is currently no clinical data on the activity of DAPD combined with MMF. This study will be the first to evaluate the addition of DAPD and MMF to a patient's current antiretroviral therapy.

At study entry, patients will be randomly assigned to one of two blinded treatment arms. Arm A receives DAPD plus MMF placebo in addition to their current regimen, while Arm B receives DAPD plus MMF in addition to their current regimen. All patients remain on their current antiretroviral regimen through Week 2. After Week 2, patients who virologically respond are encouraged to remain on blinded study treatment through Week 24. Patients who do not virologically respond are unblinded.

After unblinding, patients who were not receiving MMF may add it to their antiretroviral regimen. Response to the addition of open-label MMF is assessed after 2 weeks. Resistance to antiretroviral agents, including DAPD, will be assessed following any virologic failure occurring after Week 2. All patients have the option of optimizing their background antiretroviral regimen at Week 2, based on the results of a pre-entry resistance assay; enfuvirtide will be made available for background therapy optimization through Week 48.

Patients who are still receiving DAPD alone or DAPD plus MMF at Week 48 and who are still responding virologically may choose to continue the study drug(s) and be followed for up to an additional 48 weeks. Throughout the study, HIV-1 RNA levels, CD4 cell counts, and study drug levels will be monitored regularly. Eye exams will be done at several study visits. Only DAPD, MMF, and MMF placebo will be supplied by this study; patients must obtain the rest of their treatment regimen through their doctor. Patients who discontinue treatment before the end of study will need to come in for a follow-up visit 4 weeks after discontinuation and may need to attend future follow-up visits at 8-week intervals, as determined by the investigator.

ELIGIBILITY:
Inclusion Criteria for Step 1:

* HIV infected
* Triple-class antiretroviral treatment, as determined by the site investigator and as defined by all of the following: a) exposure to 2 or more nucleotide reverse transcriptase inhibitors (NRTIs) for at least 3 months each; b) exposure to 2 or more non-boosted protease inhibitors (PIs) for at least 3 months each, or exposure to a dual PI regimen for at least 3 months; and c) exposure to at least 1 non-nucleotide reverse transcriptase inhibitor (NNRTI) for at least 3 months.
* CD4 cell count of at least 50 cells/mm3 within 45 days prior to study entry
* Viral load of 2000 copies/ml or more within 45 days prior to study entry
* On current antiretroviral treatment regimen for at least 30 days prior to study entry. If current treatment includes abacavir, abacavir must be discontinued at least 30 days prior to study entry.
* Willing to use acceptable methods of contraception

Exclusion Criteria for Step 1:

* Pregnant or breastfeeding
* Allergy or sensitivity to the study drugs and their formulations
* Diabetes mellitus
* Cataracts or any measurable loss of vision due to lens opacity
* Best-corrected visual acuity worse than 20/200
* Certain drugs or vaccines within 30 days prior to study entry
* History of any of the following: kidney disease; serious illness within 14 days prior to study entry; end organ cytomegalovirus infection; Kaposi's sarcoma; cataracts; active herpetic infection or peptic ulcer disease within 12 months; or malabsorption, severe chronic diarrhea, or inability to eat 1 or more meals a day because of chronic nausea, emesis, or abdominal/mouth and throat discomfort
* Current alcohol or drug abuse that would interfere with adherence to study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56
Dates: Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Margolis, MD, Study Chair — Division of Infectious Diseases, University of Texas Southwestern Medical Center
Locations (17):
- United States (17):
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - UC Davis Medical Center, Sacramento, California
  - Univ. of California Davis Med. Ctr., ACTU, Sacramento, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Washington U CRS, St Louis, Missouri
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Case CRS, Cleveland, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Univ. of Pennsylvania Health System, Presbyterian Med. Ctr., Philadelphia, Pennsylvania
  - Pitt CRS, Pittsburgh, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Chapuis AG, Paolo Rizzardi G, D'Agostino C, Attinger A, Knabenhans C, Fleury S, Acha-Orbea H, Pantaleo G. Effects of mycophenolic acid on human immunodeficiency virus infection in vitro and in vivo. Nat Med. 2000 Jul;6(7):762-8. doi: 10.1038/77489. PMID 10888924
- [Background] Coull JJ, Turner D, Melby T, Betts MR, Lanier R, Margolis DM. A pilot study of the use of mycophenolate mofetil as a component of therapy for multidrug-resistant HIV-1 infection. J Acquir Immune Defic Syndr. 2001 Apr 15;26(5):423-34. doi: 10.1097/00126334-200104150-00004. PMID 11391161
- [Background] Gulick RM. New antiretroviral drugs. Clin Microbiol Infect. 2003 Mar;9(3):186-93. doi: 10.1046/j.1469-0691.2003.00570.x. PMID 12667250
- [Background] Rizzardi GP, Lazzarin A, Pantaleo G. Potential role of immune modulation in the effective long-term control of HIV-1 infection. J Biol Regul Homeost Agents. 2002 Jan-Mar;16(1):83-90. PMID 12003181